CLINICAL TRIAL: NCT02060097
Title: Effects of 24-week Cocoa Flavanol Supplementation on Photo-aged Facial Skin
Brief Title: Effects of Cocoa Flavanol on Skin Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Ho Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N0000697
Record Dates: First submitted 2014-02-09; First posted 2014-02-11 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Ageing; Photo-aging
Keywords: Anti-aging; High-flavanol cocoa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cocoa flavanol beverage (Active Comparator): flavanol 320mg/day
  Interventions: Dietary Supplement: Cocoa flavanol beverage
- Placebo beverage (Placebo Comparator): no flavanol
  Interventions: Dietary Supplement: Placebo beverage

INTERVENTIONS:
Dietary Supplement: Cocoa flavanol beverage
  Other Names: High-flavanol cocoa
  Arms: Cocoa flavanol beverage
Dietary Supplement: Placebo beverage
  Arms: Placebo beverage

SUMMARY:
Photoaging is caused by the superposition of chronic ultraviolet (UV)-induced damage on the intrinsic aging process, and accounts for the majority of age-associated changes in skin appearance. Reactive oxygen species (ROS) likely contribute to this process. Strategies utilizing endogenous skin antioxidants as well as plant-derived or synthetic compounds have been examined.

Cocoa beans fresh from the tree are exceptionally rich in polyphenols, such as flavanol, and have a higher antioxidant capacity. The present study is designed to investigate the effects of long-term intake of a product rich in cocoa flavanols on facial wrinkles, hydration, elasticity and photosensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females aged ≥ 40 years
* Facial wrinkle grade ≥ 2

Exclusion Criteria:

* received medical or cosmetic treatment that interferes with the general aging process at least 3 months before the study
* reported taking functional foods 1 month before the study
* history of acute or chronic disease such as severe liver or kidney disease or uncontrolled diabetes
* history of allergies against any component of trial foods
* any visible skin disease that might be confused with a skin reaction to the test procedure

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in skin wrinkles at week 24 | baseline, week 24
  Facial wrinkles in the crow's feet area measured as R1-3

SECONDARY OUTCOMES:
Change from baseline in skin elasticity at week 24 | baseline, week 24
  Facial elasticity measured as R2, R5, R7
Change from baseline in minimal erythema dose at week 24 | baseline, week 24
Change from baseline in skin hydration at week 12 | baseline, week 12
  Skin hydration measured by Corneometer
Change from baseline in skin color at week 12 | baseline, week 12
  Skin color measured as erythema index and melanin index

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ho Chung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Williams S, Tamburic S, Lally C. Eating chocolate can significantly protect the skin from UV light. J Cosmet Dermatol. 2009 Sep;8(3):169-73. doi: 10.1111/j.1473-2165.2009.00448.x. PMID 19735513
- [Background] Heinrich U, Neukam K, Tronnier H, Sies H, Stahl W. Long-term ingestion of high flavanol cocoa provides photoprotection against UV-induced erythema and improves skin condition in women. J Nutr. 2006 Jun;136(6):1565-9. doi: 10.1093/jn/136.6.1565. PMID 16702322
- [Derived] Yoon HS, Kim JR, Park GY, Kim JE, Lee DH, Lee KW, Chung JH. Cocoa Flavanol Supplementation Influences Skin Conditions of Photo-Aged Women: A 24-Week Double-Blind, Randomized, Controlled Trial. J Nutr. 2016 Jan;146(1):46-50. doi: 10.3945/jn.115.217711. Epub 2015 Nov 18. PMID 26581682